CLINICAL TRIAL: NCT05603143
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of GS-5245 for the Treatment of COVID-19 in Participants With High-Risk for Disease Progression
Brief Title: Study of Obeldesivir in Participants With COVID-19 Who Have a High Risk of Developing Serious or Severe Illness
Acronym: BIRCH
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was stopped early as it was determined there would not be a statistically significant treatment effect associated with the primary endpoint due to the low number of events.
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-611-6273; 2022-002741-18 (EudraCT Number)
Record Dates: First submitted 2022-10-31; First posted 2022-11-02 (Actual); Results first posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Obeldesivir (Experimental): Participants will receive obeldesivir 350 mg orally twice daily for 5 days.
  Interventions: Drug: Obeldesivir
- Placebo (Placebo Comparator): Participants will receive placebo-to-match obeldesivir orally twice daily for 5 days.
  Interventions: Drug: Obeldesivir Placebo

INTERVENTIONS:
Drug: Obeldesivir — Tablets administered orally without regard to food.
  Other Names: GS-5245
  Arms: Obeldesivir
Drug: Obeldesivir Placebo — Placebo tablets administered orally without regard to food.
  Arms: Placebo

SUMMARY:
The goal of this clinical study is to test how well the study drug, obeldesivir (GS-5245), works and how safe it is in treating coronavirus disease 2019 (COVID-19) in participants that have a higher risk of getting a serious illness.

ELIGIBILITY:
Key Inclusion Criteria:

* Willing and able to provide written informed consent.
* Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection confirmed by PCR or an approved alternative assay (eg. Rapid Antigen Test) ≤ 5 days before randomization. Serologic tests will not be accepted.
* Initial onset of COVID-19 signs/symptoms ≤ 5 days before randomization.
* Not currently hospitalized or requiring hospitalization.
* Presence of ≥ 1 risk factor (if unvaccinated) or ≥ 2 risk factors (if vaccinated at any point) for progression to severe disease.

Key Exclusion Criteria:

* Anticipated use of COVID-19 therapies during the current COVID-19 illness.
* Received any direct acting antiviral drug against SARS-CoV-2 for the treatment of COVID-19 < 28 days or < 5 half-lives, whichever is longer, before randomization.
* Anticipated need for hospitalization < 48 hours after randomization.
* New oxygen requirement < 24 hours before randomization.
* Decompensated cirrhosis (Child-Pugh class B or C) or acute liver injury/failure.
* Undergoing dialysis, or history of moderate to severe renal impairment.
* Pregnant or breastfeeding (nursing).
* Unwilling to use protocol-mandated birth control.
* Received an approved, authorized or investigational COVID-19 vaccine (including booster dose) <120 days before randomization.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 468 (Actual)
Dates: Start 2022-11-05 (Actual); Primary Completion 2023-11-07 (Actual); Study Completion 2023-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (81):
- Brazil (3):
  - Faculdade de Medicina da Universidade Federal de Minas Gerais, Belo Horizonte - MG
  - L2iP Instituto de Pesquisas Clínicas, Brasília - DF
  - Centro de Pesquisa Clinica da Universidade Municipal de São Caetano do Sul (USCS), São Caetano Do Sul - SP
- Bulgaria (18):
  - Multiprofile Hospital for Active Treatment Puls AD, Department of Internal Diseases, Blagoevgrad
  - Medical Center Asklepii OOD, Dupnitsa
  - Specialìzed Hosp¡tal for Active Trealment of Pneumophthisiatric Diseases Haskovo EOOD, Department of pneumology and phthisiatry, Haskovo
  - Medical Center Zdrave-1 OOD, Kozloduy
  - Diagnostic Consultative Center 1 - Lon EOOD, Lom
  - Medical Center Hera EOOD, Montana, Montana
  - Multiprofile Hospital for Active Treatment Dr. Stamen Iliev AD, Department of Pneumology Phthisiatrics, Montana
  - Medical Center Medconsult Pleven OOD, Pleven
  - Diagnostic Consultative Center Sveti Georgi EOOD, Plovdiv
  - MHAT Sveta Karidad EAD, First Department of Anesthesiology and Intensive Care, Plovdiv
  - Multiprofile Hospital for Active Treatment Sveti Panteleymon EOOD, First Department of Internal Diseases, Plovdiv
  - Medical Center Prolet EOOD, Rousse
  - Multiprofile Hospital for Active Treatment - Samokov EOOD, Department of Internal Diseases, Samokov
  - Medical Center Unimed EOOD, Sevlievo
  - Diagnostic and Consulting Center Aleksandrovska EOOD, Sofia
  - Medical Center Hera EOOD, Sofia
  - Diagnostic Consultative Center XX - Sofia EOOD, Sofia
  - Specialized Hospital for Active Treatment of Pneumophthisiatric Diseases-Vratsa EOOD, Department of Pneumology, Vratsa
- Canada (3):
  - Hamilton Medical Research Group, Hamilton
  - Dr. Anil K. Gupta Medicine Professional Corporation, Toronto
  - Vancouver ID Research and Care Centre Society, Vancouver
- France (2):
  - CHU de Montpellier-Hopital La Colombiere, Montpellier
  - Hopital Pitie Salpetriere, Paris
- Debreceni Egyetem Klinikai Kozpont, Debrecen, Hungary
- Unita Operativa Di Malattie Infettive Ospedale San Raffaele S.r.l., Milan, Italy
- Japan (3):
  - IUHW Narita Hospital, Chibaken
  - Okayama University Hospital, Okayama
  - Suita Municipal Hospital, Suita
- Mexico (8):
  - Panamerican Clinical Research Mexico S.A. de C.V., Col. El Salitre Juriquilla
  - Neurociencias Estudios Clinicos S.C., Culiacan Sinaloa
  - PanAmerican Clinical Research Mexico S.A de C.V., Guadalajara
  - Clinstile, S.A. De C.V., Mexico City
  - EME RED Hospitalaria, Mérida
  - Kohler & Milstein Research S.A de C.V., Mérida
  - Oaxaca Site Management Organization S.C., Oaxaca City
  - FAICIC S. de R.L. de C.V., Veracruz
- Poland (3):
  - Ginemedica OVO 21, Wroclaw
  - ETG Lodz, Zgierz
  - ClinMedica Research, Skierniewice, Łódź Voivodeship
- Portugal (3):
  - Hospital CUF Descobertas, Lisbon
  - Centro Hospitalar de Entre Douro e Vouga - Hospital de Sao Sebaststiao, Santa Maria da Feira
  - Hospital da Luz - Arrabida, Vila Nova de Gaia
- Romania (3):
  - "Prof. Dr. Matei Bals" National Institute for Infectious Diseases, Bucharest
  - County Hospital Caracal, Caracal
  - Sibiu Emergency Clinical County Hospital, Sibiu
- National Centre for Infectious Diseases, Tan Tock Seng Hospital, Singapore, Singapore
- South Africa (8):
  - Madibeng Centre for Research, Brits
  - Clinresco Centres (Pty) Ltd, City of Johannesburg
  - Synapta Clinical Research Centre, Durban
  - Perinatal HIV Research Unit (PHRU), Johannesburg
  - Global Clinical Trials, Pretoria
  - Jongaie Research, Pretoria West
  - Limpopo Clinical Research Initiative, Thabazimbi
  - FCRN Clinical Trial Centre (Pty) Ltd, Vereeniging
- South Korea (3):
  - ChungNam National University Hospital, Daejeon
  - Chonnam National University Bitgoeul Hospital, Gwangju
  - Korea University Guro Hospital, Seoul
- Spain (12):
  - Hospital Universitario Virgen de Las Nieves., A Gudiña
  - Hospital General Universitario Dr. Balmis, Alicante
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - CAP La Mina, Barcelona
  - Hospital HM Nou Delfos, Barcelona
  - Hospital Universitario Virgen del Rocio, Las Cabezas de San Juan
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Puerta de Hierro - Majadahonda, Majadahonda
  - Hospital General Universitario Reina Sofia, Murcia
  - Hospital Universitario Son Espases, Palma de Mallorca
  - Hospital Universitaro y Politecnico La Fe, Valencia
- Taiwan (5):
  - Hualien Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation, Hualien City
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Tao-Yuan General Hospital, Taoyuan
  - Kaohsiung Veterans General Hospital, Zuo Ying Qu
- Acibadem University School of Medicine Atakent Hospital, Trabzon, Turkey (Türkiye)
- United Kingdom (3):
  - Ormeau Clinical Trials Limited, Belfast
  - Lakeside Healthcare, Corby
  - CPS Research, Glasgow

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hedskog C, Rodriguez L, Hu Y, Li J, Han D, Peinovich N, Martinez C, Ho PY, Perry JK, Del Castillo JMG, Koullias Y, Martin R, Hyland RH. SARS-CoV-2 Resistance Analyses From the Phase 3 BIRCH Study of Obeldesivir in High-Risk Nonhospitalized Participants With COVID-19. Antiviral Res. 2026 Jan 19:106351. doi: 10.1016/j.antiviral.2026.106351. Online ahead of print. PMID 41565160
- [Derived] Streinu-Cercel A, Castagna A, Chang SC, Chen YS, Koullias Y, Mozaffarian A, Hyland RH, Humeniuk R, Caro L, Davies S, Rodriguez L, Hedskog C, Chen S, Etchevers K, Behenna-Renton N, Llewellyn J, Osinusi A, Duff F, Barrat Hernandez A, McNally D, Simon-Campos JA, Leal FE, Fouche LF, Gonzalez Del Castillo JM. Efficacy and Safety of Obeldesivir in High-Risk Nonhospitalized Patients With COVID-19 (BIRCH): A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study. Clin Infect Dis. 2026 Feb 9;82(1):e24-e32. doi: 10.1093/cid/ciaf406. PMID 40694627
- See also: Gilead Clinical Trials Website — http://www.gileadclinicaltrials.com/study/?id=GS-US-611-6273

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the South America, Europe, North America, Africa and Asia.
Pre-assignment Details: 515 participants were screened.
Groups:
- Obeldesivir: Participants received obeldesivir 350 mg orally twice daily for 5 days.
- Placebo: Participants received placebo-to-match obeldesivir orally twice daily for 5 days.
Period: Overall Study
Arm/Group | Obeldesivir | Placebo
Started | 233 | 235
Completed | 224 | 227
Not Completed | 9 | 8
Not completed — Withdrew consent | 6 | 2
Not completed — Randomized but never treated | 0 | 3
Not completed — Adverse Event | 2 | 0
Not completed — Death | 0 | 1
Not completed — Investigator's discretion | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: The All Randomized Analysis Set included all participants who were randomized in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Obeldesivir | Placebo | Total
Number analyzed (Participants) | 233 | 235 | 468
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (14.9) | 53 (16.6) | 55 (15.8)
Age, Customized [Count of Participants; unit: Participants]
  Adults (18 - 64 Years) | 159 | 173 | 332
  Geriatrics (65 - 84 Years) | 71 | 59 | 130
  Geriatrics (85 Years and Over) | 3 | 3 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 147 | 117 | 264
  Male | 86 | 118 | 204
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 36 | 43 | 79
  Not Hispanic or Latino | 197 | 192 | 389
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 178 | 168 | 346
  Asian | 24 | 32 | 56
  American Indian or Alaska Native | 21 | 19 | 40
  Black or African American | 9 | 10 | 19
  Other or More Than One Race | 1 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Romania | 29 | 24 | 53
  Singapore | 1 | 0 | 1
  Hungary | 0 | 1 | 1
  Japan | 2 | 3 | 5
  United Kingdom | 8 | 0 | 8
  Portugal | 4 | 5 | 9
  Spain | 11 | 12 | 23
  Canada | 7 | 11 | 18
  South Korea | 1 | 2 | 3
  Turkey | 1 | 1 | 2
  Taiwan | 17 | 23 | 40
  Brazil | 3 | 5 | 8
  Poland | 12 | 7 | 19
  Italy | 1 | 1 | 2
  Mexico | 24 | 24 | 48
  South Africa | 15 | 16 | 31
  Bulgaria | 97 | 99 | 196
  France | 0 | 1 | 1
Baseline Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Nasal Swab Viral Load [Mean (Standard Deviation); unit: log10 copies/mL] — Population: The Safety Analysis Set included all participants who received at least 1 dose of study drug with data available were analyzed. One participant randomized to placebo arm received obeldesivir and was counted in obeldesivir group for the analysis of this baseline measure.
  log10 copies/mL
    number analyzed (Participants) | 218 | 215 | 433
    (all) | 6.15 (1.629) | 6.15 (1.622) | 6.15 (1.624)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Coronavirus Disease 2019 (COVID-19) Related Hospitalization or All-Cause Death by Day 29
Description: COVID-19-related hospitalization was defined as ≥ 24 hours of acute care for a reason related to COVID-19, in a hospital or similar acute care facility, including emergency rooms or temporary facilities instituted to address medical needs of those with COVID-19. This included specialized acute medical care units within an assisted living facility or nursing home. This did not include hospitalization for the purposes of public health and/or clinical trial execution. The date and duration of hospital admission, and primary reason for hospitalization (including if the hospitalization was related to COVID-19) were recorded. Percentages were rounded off.
Time Frame: Up to Day 29
Population: The Full Analysis Positive Set included all randomized participants who received at least 1 dose of study drug and were SARS-CoV-2 positive at baseline as confirmed by cepheid's xpert xpress coronavirus-2/flu/respiratory syncytial virus plus test or SARS-CoV-2 reverse transcriptase quantitative polymerase chain reaction test from the central laboratory.
Measure: Number; unit: percentage of participants
Arm/Group | Obeldesivir | Placebo
Number analyzed (Participants) | 211 | 207
percentage of participants | 0 | 0.5
Statistical Analysis 1: Comparison: Obeldesivir vs Placebo; Test type: Other; p = 0.3161, Log Rank

2. Secondary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAE)
Description: TEAEs were defined as 1 or both of the following:
  Any AEs with an onset date on or after the study drug start date and no later than 30 days after permanent discontinuation of study drug. Any AEs leading to premature discontinuation of study drug. Percentages were rounded off.
Time Frame: First dose date up to 5 Days plus 30 Days
Population: The Safety Analysis Set included all participants who received at least 1 dose of study drug. One participant randomized to placebo arm received obeldesivir and was counted in obeldesivir group for the analysis of this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Obeldesivir | Placebo
Number analyzed (Participants) | 234 | 231
percentage of participants | 22.2 | 20.8

3. Secondary Outcome: Percentage of Participants Experiencing Laboratory Abnormalities
Description: Treatment-emergent laboratory abnormalities were defined as values that increase at least 1 toxicity grade from baseline at any postbaseline time point, up to and including the date of last dose of study drug plus 30 days. Percentages were rounded off.
Time Frame: First dose date up to 5 Days plus 30 Days
Population: Participants from the Safety Analysis Set who had available post baseline data were analyzed. One participant randomized to placebo arm received obeldesivir and was counted in obeldesivir group for the analysis of this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Obeldesivir | Placebo
Number analyzed (Participants) | 230 | 227
percentage of participants
  Any grade | 56.1 | 61.7
  Grade 3 or 4 | 6.5 | 4.8

4. Secondary Outcome: Percentage of Participants Experiencing Serious Adverse Events (SAEs) and Adverse Events (AEs) Leading to Study Drug Discontinuation
Description: A treatment emergent AE is defined as an AE that occurs or worsens in severity on or after the date of the first dose of study drug but no later than 30 days after the permanent discontinuation of study drug or an AE leading to discontinuation of study drug. A SAE is defined as an event that, at any dose, resulted in any of the following: death, life-threatening, in-patient hospitalization or prolongation of existing hospitalization, persistent or significant disability/incapacity, a congenital anomaly/birth defect, or a medically important event or reaction. Percentages were rounded off.
Time Frame: First dose date up to 5 Days plus 30 Days
Population: Participants in the Safety Analysis Set were analyzed. One participant randomized to placebo arm received obeldesivir and was counted in obeldesivir group for the analysis of this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Obeldesivir | Placebo
Number analyzed (Participants) | 234 | 231
percentage of participants
  AEs Leading to Study Drug Discontinuation | 1.7 | 0.9
  SAEs Leading to Study Drug Discontinuation | 0.9 | 0.9

5. Secondary Outcome: Percentage of Participants With All-Cause Hospitalization by Day 29
Description: All-cause hospitalization was defined as ≥ 24 hours of acute care, in a hospital or similar acute care facility, including emergency rooms or temporary facilities instituted to address medical needs of those with COVID-19. This includes specialized acute medical care units within an assisted living facility or nursing home. This does not include hospitalization for the purposes of public health and/or clinical study execution. The date and duration of hospital admission, and primary reason for hospitalization (including if the hospitalization is related to COVID-19) were recorded. Percentages were rounded off.
Time Frame: Up to Day 29
Population: Participants in the Full Analysis Positive Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Obeldesivir | Placebo
Number analyzed (Participants) | 211 | 207
percentage of participants | 0.5 | 0
Statistical Analysis 1: Comparison: Obeldesivir vs Placebo; Test type: Other; p = 0.3219, Log Rank

6. Secondary Outcome: Percentage of Participants With COVID-19-Related Medically Attended Visits (MAVs) or All-Cause Death by Day 29
Description: Medically attended visits were defined as interactions with health care professionals other than study staff or designees including hospitalization; in-person emergency, urgent, or primary care visits; or any other in-person visit attended by the participant and a health care professional. The nature and cause of the visit were identified. KM estimates were used in the outcome measure analysis. Percentages were rounded off.
Time Frame: Up to Day 29
Population: Participants in the Full Analysis Positive Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Obeldesivir | Placebo
Number analyzed (Participants) | 211 | 207
percentage of participants | 1.0 | 1.0
Statistical Analysis 1: Comparison: Obeldesivir vs Placebo; Test type: Other; p = 0.6568, Log Rank; Hazard Ratio (HR) = 1.496, 95% CI 2-sided [0.250 to 8.952] — Hazard ratio and two-sided 95% CI for hazard ratio were estimated using the Cox regression

7. Secondary Outcome: Percentage of Participants With COVID-19-Related MAVs by Day 29
Description: as for outcome 6
Time Frame: Up to Day 29
Population: Participants in the Full Analysis Positive Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Obeldesivir | Placebo
Number analyzed (Participants) | 211 | 207
percentage of participants | 1 | 0.5
Statistical Analysis 1: Comparison: Obeldesivir vs Placebo; Test type: Other; p = 0.3190, Log Rank; Hazard Ratio (HR) = 2.990, 95% CI 2-sided [0.311 to 28.740] — Hazard ratio and two-sided 95% CI for hazard ratio were estimated using the Cox regression

8. Secondary Outcome: Percentage of Participants With All-cause Death by Day 29
Description: Percentages were rounded off.
Time Frame: Up to Day 29
Population: Participants in the Full Analysis Positive Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Obeldesivir | Placebo
Number analyzed (Participants) | 211 | 207
percentage of participants | 0 | 0.5
Statistical Analysis 1: Comparison: Obeldesivir vs Placebo; Test type: Other; p = 0.3161, Log Rank

9. Secondary Outcome: Time to COVID-19 Symptom Alleviation by Day 15
Description: Time to COVID-19 symptom alleviation was calculated as symptom alleviation date/time minus the first dose date/time. Symptom alleviation was evaluated for the 15 targeted symptoms using symptoms of infection with coronavirus-19 (SIC) questionnaire. The SIC questionnaire assessed all targeted symptoms, alleviation was defined as the SIC rating of 0, or at least 3 points decrease in rating from baseline, or an answer "No" to the question for at least 48 consecutive hours.
Time Frame: Up to Day 15
Population: Participants in the Full Analysis Positive Set with Covid19 symptoms who completed Symptoms of Infection With Coronavirus-19 at baseline were analyzed.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Obeldesivir | Placebo
Number analyzed (Participants) | 84 | 78
Days | 7.3 [5.4 to 9.4] | 9.3 [6.5 to NA] — Upper limit of CI did not reach due to low number of participants with events.
Statistical Analysis 1: Comparison: Obeldesivir vs Placebo; Test type: Other; p = 0.0859, Log Rank — P-value was based on stratified Log-rank test with randomization stratification factors as the strata; Hazard Ratio (HR) = 1.425, 95% CI 2-sided [0.961 to 2.112] — Hazard ratio and two-sided 95% CI for hazard ratio were estimated using the Cox regression with randomization stratification factors as covariates

10. Secondary Outcome: Change From Baseline in Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Nasal Swab Viral Load at Day 5
Description: The mixed model for repeated measures (MMRM) was used for analysis.
Time Frame: Day 5
Population: Virology Analysis Set included all randomized participants who received at least 1 dose of study drug and had baseline SARS-CoV-2 viral load greater than or equal to lower limit of quantitation.
Measure: Least Squares Mean (Standard Error); unit: log10 copies/mL
Arm/Group | Obeldesivir | Placebo
Number analyzed (Participants) | 193 | 192
log10 copies/mL | -2.80 (0.092) | -2.22 (0.092)
Statistical Analysis 1: Comparison: Obeldesivir vs Placebo; Test type: Other; p < 0.0001, MMRM; Treatment Difference (vs Placebo) = -0.58, 95% CI 2-sided [-0.83 to -0.33] — Least-squares mean (SE), 95% CI and P value were from MMRM with baseline viral load and randomization strata as covariates

11. Secondary Outcome: Plasma Concentrations of GS-441524 (Metabolite of Obeldesivir)
Time Frame: Day 1, 0.75 and 2 hours postdose and Day 5 predose and 0.75 hours postdose
Population: Pharmacokinetic Analysis Set included all randomized participants who received at least 1 dose of study drug and had at least 1 non missing concentration value reported by the PK laboratory with available data were analyzed .
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Obeldesivir
Number analyzed (Participants) | 224
ng/mL
  Day 1, 0.75 hours postdose: number analyzed (Participants) | 216
  Day 1, 0.75 hours postdose | 2330.42 (1709.560)
  Day 1, 2 hours postdose: number analyzed (Participants) | 95
  Day 1, 2 hours postdose | 2535.84 (1370.131)
  Day 5, Predose: number analyzed (Participants) | 170
  Day 5, Predose | 1116.81 (1101.371)
  Day 5, 0.75 hours postdose: number analyzed (Participants) | 174
  Day 5, 0.75 hours postdose | 3089.09 (1839.992)

ADVERSE EVENTS:
Time Frame: All-cause mortality, Adverse events: First dose date up to 5 Days plus 30 Days
Description: All-cause mortality: All Randomized Analysis Set included all participants who were randomized in the study. One participant randomized to placebo arm accidentally received obeldesivir and was counted in obeldesivir group for the analysis of all-cause mortality and adverse events.
  Adverse events: Safety Analysis Set included all participants who were randomized and received at least 1 dose of study drug.
Arm/Group | Obeldesivir | Placebo
All-Cause Mortality (participants affected / at risk) | 0/234 | 1/234
Serious Adverse Events (participants affected / at risk) | 2/234 | 2/231
Other Adverse Events (participants affected / at risk) | 0/234 | 0/231
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Obeldesivir (N=234) | Placebo (N=231)
Vomiting (Gastrointestinal disorders) | 0 | 1
Death (General disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2023-03-29): https://cdn.clinicaltrials.gov/large-docs/43/NCT05603143/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-22): https://cdn.clinicaltrials.gov/large-docs/43/NCT05603143/SAP_001.pdf